CLINICAL TRIAL: NCT02811939
Title: Testing the Interactive Effects of Delta-9-Tetrahydrocannabinol and Pregnenolone: Sub-Study I
Acronym: THC-PREG-I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1501015242.A
Record Dates: First submitted 2016-03-15; First posted 2016-06-23 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Healthy
Keywords: Cannabis; Marijuana; THC; Dronabinol; Pregnenolone; PREG; Psychotic Disorders
MeSH Terms: conditions — Marijuana Abuse; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active THC and Placebo Pregnenolone (Experimental)
  Interventions: Drug: Active Dronabinol; Drug: Placebo Pregnenolone
- Active THC and Active Pregnenolone (Experimental)
  Interventions: Drug: Active Dronabinol; Drug: Active Pregnenolone
- Placebo THC and Active Pregnenolone (Experimental)
  Interventions: Drug: Active Pregnenolone; Drug: Placebo Dronabinol
- Placebo THC and Placebo Pregnenolone (Placebo Comparator)
  Interventions: Drug: Placebo Dronabinol; Drug: Placebo Pregnenolone

INTERVENTIONS:
Drug: Active Dronabinol — 20 mg capsule of Dronabinol will be administered orally
  Arms: Active THC and Active Pregnenolone; Active THC and Placebo Pregnenolone
Drug: Active Pregnenolone — 1.79 mg/kg of Pregnenolone will be administered sublingually (under the tongue)
  Arms: Active THC and Active Pregnenolone; Placebo THC and Active Pregnenolone
Drug: Placebo Dronabinol — Control: Placebo pill (no active cannabinoids) administered orally
  Arms: Placebo THC and Active Pregnenolone; Placebo THC and Placebo Pregnenolone
Drug: Placebo Pregnenolone — Control: Placebo given sublingually (under the tongue)
  Arms: Active THC and Placebo Pregnenolone; Placebo THC and Placebo Pregnenolone

SUMMARY:
The overall purpose of this study is to examine the effect of Pregnenolone (PREG) on the acute psychosis-like and cognitive effects of Delta-9-Tetrahydrocannabinol (THC). This will be tested by pretreating healthy individuals with PREG, and then assessing their responses to Dronabinol (THC).

ELIGIBILITY:
Inclusion Criteria:

* Exposed to cannabis at least once in lifetime

Exclusion Criteria:

* Cannabis naïve
* Individuals with a documented reaction/allergy to Pregnenolone
* Individuals with a documented reaction/allergy to Sesame oil

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-06-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline: Positive and Negative Syndrome Scale (PANSS) | baseline, 30, 110, 180, and 240 minutes after the administration of oral dronabinol/placebo
  Positive, negative and general symptoms will be assessed using the positive, negative, and general symptom subscale of the PANSS.

SECONDARY OUTCOMES:
Change from Baseline: Clinician Administered Dissociative Symptoms Scale (CADSS) | baseline, 30, 110, 180, and 240 minutes after the administration of oral dronabinol/placebo
  Perceptual alterations will be measured using the CADSS. This is a scale consisting of 19 self-reported items, and 9 clinician-rated items. The scale captures alterations in environmental/time/body perception, feelings of unreality, and memory impairment.
Change from Baseline: Visual Analog Scale (VAS) | Baseline; 30 minutes and 10 minutes prior to administration of oral dronabinol or placebo; 20, 90, 110, 150, 180, and 240 minutes after the administration of oral dronabinol/placebo
  Feeling states associated with cannabis intoxication will be measured using a self-reported visual analog scale of feeling states associated with cannabis effects (ex. "high, "calm", "anxious"). Subjects will be asked to score the perceived intensity of these feeling states at that moment on a 11mm line. This data will be captured to validate the experiment is relevant to cannabis effect.
Change from Baseline: Psychotomimetic States Inventory (PSI) | baseline, 30, 110, 180, and 240 minutes after the administration of oral dronabinol/placebo
  The PSI is a measure of drug induced psychotomimetic states. This self-reported scale consists of 28 items rated 0 (not at all) to 3 (extremely) and will facilitate the characterization of a wide range of dissociative/hallucinatory phenomena as well as cognitive disorganization associated with the administration of THC.
Cognitive Test Battery | 25 minutes after Dronabinol is given orally
  Several computer tasks will be administered in order to evaluate the effects of cannabis on verbal learning and memory. The battery consists of five computer tasks that last no longer than 20 minutes in total.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Cyril D'Souza, MD, Principal Investigator — Yale Univerisity, School of Medicine
Locations (1):
- Biological Studies Unit at the VA Connecticut Healthcare System, Yale School of Medicine, West Haven, Connecticut, United States